CLINICAL TRIAL: NCT03145883
Title: Effects of Aerobic Exercise on Asthmatic Responses in Obese Adults
Brief Title: Exercise and Asthma in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Arizona Biomedical Research Commission (ABRC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1504818055
Record Dates: First submitted 2017-05-01; First posted 2017-05-09 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-04

CONDITIONS: Asthma in Overweight Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group
- Home-based Aerobic Exercise (Experimental): Participants will be prescribed weekly exercise goals starting with 75 minutes a week (e.g., 15 minutes per day, 5 days a week) and progressed to 200 minutes a week (e.g., 40 minutes per day, 5 days a week) by week 12. Exercise will consist of participant preference of mobility exercises, most likely walking. Aerobic exercise, similar to a brisk walk, will be recommended as the primary mode of exercise.
  Interventions: Other: Home-Based Aerobic Exercise

INTERVENTIONS:
Other: Home-Based Aerobic Exercise
  Arms: Home-based Aerobic Exercise

SUMMARY:
This pilot study will use an unmasked, parallel group, randomized design. Thirty adult overweight or obese subjects with mild-moderate persistent asthma will be randomly assigned to one of two groups: 12-weeks of home-based moderate intensity aerobic exercise versus no intervention. The study will include 2 clinic visits and 12 telephone calls. Exercise testing to assess physical fitness levels will occur during visits 1 and 2. Blood sampling for biomarkers, inflammatory markers, and other assessments will be done.

DETAILED DESCRIPTION:
The primary aim of this pilot study is to recruit and retain obese adults with mild-moderate persistent asthma for a study protocol that includes exercise at a moderate intensity level in a home-based setting. The investigators primary hypothesis is that compared to no intervention, 12-weeks of moderate intensity aerobic exercise will attenuate serum levels of adipokines (leptin, adiponectin), and other pro-inflammatory markers. The investigators will also analyze the effect of the intervention on fitness levels, pulmonary function, asthma symptoms, asthma control, and asthma-related quality of life.

Given that this is a proof of concept/feasibility study, there is no primary outcome measure. The following measures will be assessed:

* Obesity related biomarkers and other markers of inflammatory responses:
* Asthma symptoms and asthma control measures:
* Lung function
* Fitness levels and physical activity levels:

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma
* Currently prescribed a daily controller asthma medication as evidence of mild-moderate persistent asthma
* Body Mass Index BMI ≥ 30-45 kg/m2

Exclusion Criteria:

* Individuals who undergo aerobic exercise regularly (3 or more times per week for more than 20 minutes) 6 months prior to the study
* Participants with very severe obesity (WHO obese class III) - BMI≥ 45 kg/m2
* Individuals with other clinically significant major illnesses, such as congenital heart disease, juvenile arthritis, inflammatory bowel disease, cystic fibrosis, or other conditions that would limit participation in the exercise protocol or interfere with study measurements will not be eligible.
* Uncontrolled hypertension (resting systolic blood pressure > 150mmHg, and/or diastolic blood pressure >90 mmHg despite anti-hypertension medications.
* Current use of beta blockers
* Currently pregnant, pregnant during the previous six months, or planning to become pregnant in the next three months as obtained by self-report.
* Participants who have experienced a clinically significant exacerbation within the past 6 weeks will be excluded. This includes an unscheduled physician visit, emergency room visit, or hospitalization related or use of systemic corticosteroids for asthma.
* Unable or unwilling to provide consent
* Unable or unwilling to perform the exercise protocol and provide study measurements,
* Inability to perform baseline measurements
* Intend to move out of the area within 3 months from the start of the study
* Inability to be contacted by telephone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Obesity related biomarkers | change from Visit 1 (baseline) and Visit 2 (end of study - 12 weeks later)
  Obesity markers will be evaluated in peripheral blood: Leptin and adiponectin, two adipokines that have been previously implicated in the link between asthma and obesity will be measured in peripheral blood via ELISA
Asthma symptoms | change from Visit 1 (baseline) and Visit 2 (end of study - 12 weeks later)
  Asthma symptoms will be measured with the Asthma Symptom Utility Index (ASUI)
Lung function | change from Visit 1 (baseline) and Visit 2 (end of study - 12 weeks later)
  Lung function will be evaluated via spirometry according to ATS guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Chrstian Bime, MD, Principal Investigator — University of Arizona, College of Medicine
Locations (1):
- The University of Arizona and the Tucson Unified School District, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No